CLINICAL TRIAL: NCT04276493
Title: Phase 1b/2 Study Investigating Safety, Tolerability, Pharmacokinetics and Preliminary Antitumor Activity of Anti-HER2 Bispecific Antibody ZW25 in Combination With Chemotherapy With/Without Tislelizumab in Patients With Advanced HER2-positive Breast Cancer or Gastric/Gastroesophageal Junction Adenocarcinoma
Brief Title: Anti-HER2 Bispecific Antibody Zanidatamab (ZW25) Activity in Combination With Chemotherapy With/Without Tislelizumab
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGB-A317-ZW25-101; CTR20210237 (Other: ChinaDrugTrials)
Record Dates: First submitted 2020-02-04; First posted 2020-02-19 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer; Gastric Cancer; Gastroesophageal Junction Cancer
MeSH Terms: conditions — Breast Neoplasms; Stomach Neoplasms | interventions — zanidatamab; Docetaxel; tislelizumab; Capecitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cohort 1- Zanidatamab + Docetaxel (Experimental): Zanidatamab intravenous (IV) infusion followed by docetaxel IV infusion first-line therapy once every three weeks (Q3W) in female participants with metastatic breast cancer
  Interventions: Biological: Zanidatamab; Drug: Docetaxel
- Cohort 2- Zanidatamab + Tiselizumab + Chemotherapy (Experimental): Zanidatamab intravenous (IV) infusion followed by tislelizumab IV infusion and CAPOX chemotherapy (oral capecitabine + IV oxaliplatin) first-line therapy once every three weeks (Q3W) in participants with metastatic gastric / GEJ adenocarcinoma
  Interventions: Biological: Zanidatamab; Biological: Tislelizumab; Drug: Capecitabine; Drug: Oxaliplatin

INTERVENTIONS:
Biological: Zanidatamab — Administered intravenously
  Other Names: ZW25
Drug: Docetaxel — Administered intravenously
  Arms: Cohort 1- Zanidatamab + Docetaxel
Biological: Tislelizumab — Administered intravenously
  Other Names: BGB-A317
  Arms: Cohort 2- Zanidatamab + Tiselizumab + Chemotherapy
Drug: Capecitabine — Administered orally
  Arms: Cohort 2- Zanidatamab + Tiselizumab + Chemotherapy
Drug: Oxaliplatin — Administered intravenously
  Arms: Cohort 2- Zanidatamab + Tiselizumab + Chemotherapy

SUMMARY:
The purpose of the study is to assess the safety, tolerability and preliminary antitumor activity of zanidatamab in combination with docetaxel in participants with human epidermal growth factor receptor 2 (HER2)-positive breast cancer, and zanidatamab in combination with tislelizumab and chemotherapy in participants with HER2-positive gastric/gastroesophageal Junction (GEJ) adenocarcinoma

ELIGIBILITY:
Key Inclusion Criteria:

1. Disease diagnosis and prior treatment:

   1. Cohort 1 (the first-line breast cancer treatment cohort):

      * Female participants with histologically or cytologically confirmed unresectable, locally advanced, recurrent or metastatic adenocarcinoma of the breast and candidate for chemotherapy. Locally recurrent disease must not be amenable to resection with curative intent.
      * Human epidermal growth factor receptor 2 (HER2) IHC 3+ or in situ hybridization positive on the archival tumor tissue or fresh biopsy sample.
      * Have not received previous systemic anticancer therapy for locally advanced unresectable or metastatic disease.
   2. Cohort 2 (the first-line gastric/gastroesophageal junction adenocarcinoma treatment cohort):

      * Histologically or cytologically confirmed unresectable, locally advanced, recurrent or metastatic adenocarcinoma of the stomach or gastroesophageal junction
      * HER2 IHC 3+ or HER2 IHC 2+ together with in situ hybridization positive on the archival tumor tissue or fresh biopsy sample.
      * Have not received previous systemic anticancer therapy for locally advanced unresectable or metastatic disease, including any approved or investigational estimated glomerular filtration rate (EGFR) or anti-HER2 agents or vaccines, cytotoxic chemotherapy or checkpoint inhibitors
2. At least 1 measurable lesion as defined per RECIST Version 1.1
3. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 1
4. Adequate organ function
5. Left ventricular ejection fraction (LVEF) ≥ 50% at baseline as determined by either echocardiogram or multigated acquisition scan (MUGA) (echocardiogram is the preferred method) within 28 days before the first dose of study drug

Key Exclusion Criteria:

1. Prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2 or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways
2. History of approved or investigative tyrosine kinase/HER inhibitors in any treatment setting

   a. except trastuzumab with or without pertuzumab used in neoadjuvant or adjuvant setting for Cohort 1
3. Active leptomeningeal disease, untreated or uncontrolled brain metastasis
4. Any active malignancy ≤ 2 years before the first dose of study drug, except for the specific cancer under investigation in this trial and any localized cancer that has been treated curatively (eg, resected basal or squamous cell skin cancer, superficial bladder cancer, carcinoma in situ of the cervix)
5. Any condition that required systemic treatment with either corticosteroids (> 10 mg daily of prednisone or equivalent) or other immunosuppressive medication ≤ 14 days before the first dose of study drug

Note: Participants who are currently or have previously been on any of the following steroid regimens are not excluded:

1. Adrenal replacement steroid (dose ≤ 10 mg daily of prednisone or equivalent)
2. Topical, ocular, intra-articular, intranasal, or inhaled corticosteroid with minimal systemic absorption
3. Short course (≤ 7 days) of corticosteroid prescribed prophylactically (eg, for contrast dye allergy) or for the treatment of a non-autoimmune condition (eg, delayed-type hypersensitivity reaction caused by contact allergen)

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2020-03-26 (Actual); Primary Completion 2023-12-07 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Number of Participants experiencing Adverse Events (AEs) | From the first dose of study drug(s) to 30 days after the last dose; up to approximately 41 months
Number of Participants experiencing Serious Adverse Events (SAEs) as assessed by the investigator. | From the first dose of study drug(s) to 30 days after the last dose; up to approximately 41 months
Objective response rate (ORR) | From the start date of study treatment to the first documentation of progression or death, whichever occurs first, up to approximately 41 months
  Defined as the percentage of participants who had a best overall response of complete response or partial response per the Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1.

SECONDARY OUTCOMES:
Duration of response (DOR) | From the start date of study treatment to the first documentation of progression or death, whichever occurs first, up to approximately 41 months
Time to response (TTR) | From the start date of study treatment to the first documentation of progression or death, whichever occurs first, up to approximately 41 months
  Time from the start date of study drug to the first determination of an objective response by investigator per RECIST Version 1.1
Progression-free survival (PFS) | From the start date of study treatment to the first documentation of progression or death, whichever occurs first, up to approximately 41 months
  Percentage of participants with best overall response of complete response, partial response, and stable disease by investigator per RECIST Version 1.1
Overall survival (OS) | From the start date of study treatment to the documented death date or the last known alive date, up to approximately 41 months
  Time from the start date of study drug to the date of death due to any cause
Serum concentration of zanidatamab as a function of time | Predose and immediately postdose
Observed maximum plasma concentration of zanidatamab during a sample interval (Cmax) | Predose and immediately postdose
Observed time to maximum plasma concentration of zanidatamab during a sampling interval (tmax) | Predose and immediately postdose
Terminal elimination half-life (t1/2) of zanidatamab | Predose and immediately postdose
Area under the plasma concentration-time curve from time zero to the last measurable timepoint (AUC(0-t)) of zanidatamab | Predose and immediately postdose
Apparent clearance after oral administration (CL/F) of zanidatamab | Predose and immediately postdose
Presence of anti-zanidatamab-antibodies | Predose and immediately postdose
Presence of zanidatamab neutralizing antibodies | Predose and immediately postdose
Number of participants with AEs and SAEs who entered the long-term extension period | From the first dose of study drug(s) to 30 days after the last dose; up to approximately 51 months

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeiGene
Locations (21):
- China (8):
  - The Affiliated Hospital of Military Medical Sciences, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Chongqing Cancer Hospital, Chongqing, Chongqing Municipality
  - Guangdong Provincial Peoples Hospital Huifu Branch, Guangzhou, Guangdong
  - The Third Hospital of Nanchang, Nanchang, Jiangxi
  - Jilin Cancer Hospital, Changchun, Jilin
  - Liaoning Cancer Hospital and Institute, Shenyang, Liaoning
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
- South Korea (8):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul, Seoul Teugbyeolsi
  - Severance Hospital Yonsei University Health System, Seoul, Seoul Teugbyeolsi
  - Asan Medical Center, Seoul, Seoul Teugbyeolsi
  - Gangnam Severance Hospital, Yonsei University Health System, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center, Seoul, Seoul Teugbyeolsi
  - Korea University Guro Hospital, Seoul, Seoul Teugbyeolsi
- Taiwan (5):
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital East Campus, Taipei
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Yes